CLINICAL TRIAL: NCT03685045
Title: Enhancing Treatment of Hepatitis C in Opioid Substitution Settings II (ETHOS II): A Partnership Project to Enhance Hepatitis C Care in Drug and Alcohol Clinics
Brief Title: ETHOS ENGAGE: Enhancing Treatment of Hepatitis C in Opioid Substitution Settings
Acronym: ETHOS II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VHCRP1509
Record Dates: First submitted 2018-09-20; First posted 2018-09-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hepatitis C
Keywords: hepatitis c; opioid substitution settings; OST; people who inject drugs; direct-acting antiviral treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: The intervention is the campaign days where all participants will undergo a questionnaire, point of care and dried blood spot testing for hepatitis C, fibroscan and a clinical assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Campaign Days (Experimental): All participants have the intervention of the campaign days which include hepatitis C screening, fibroscans and clinical assessments.
  Interventions: Procedure: Campaign days

INTERVENTIONS:
Procedure: Campaign days — Participants who consent will complete study procedures (Hep C test, fibroscan, questionnaire, clinical assessment) and followed up through medical record review.

SUMMARY:
The overall goals of the ETHOS II Project are to enhance hepatitis C virus (HCV) care in drug treatment clinics and needle and syringe programs (NSPs) in New South Wales and Australia, and to develop a translational framework for subsequent establishment of HCV screening and treatment programs in drug treatment clinics and NSPs across NSW and nationally.

DETAILED DESCRIPTION:
The ETHOS II Project is a collaborative research project led by the Kirby Institute, UNSW Sydney, in partnership with:

* The Centre for Social Research in Health, UNSW Sydney
* NSW Health
* NSW Users and AIDS Association
* Hepatitis NSW
* Australasian Society for HIV, Viral Hepatitis and Sexual Health Medicine (ASHM)

The overall goals of the ETHOS II Project are to enhance hepatitis C virus (HCV) care in drug treatment clinics and needle and syringe programs (NSPs) in New South Wales and Australia, and to develop a translational framework for subsequent establishment of HCV screening and treatment programs in drug treatment clinics and NSPs across NSW and nationally.

The ETHOS II Project is divided into three parts:

I. ETHOS ENGAGE cohort; II. Qualitative research on barriers/facilitators to HCV care; III. HCV toolkit, education and training.

Part I: ETHOS ENGAGE The ETHOS ENGAGE cohort is a non-randomised trial to assess the effect of an intervention incorporating on-site HCV RNA testing, liver fibrosis assessment, and linkage to care to enhance scale-up of direct-acting antiviral therapy for HCV infection among people with a history of injecting drug use, and recent injecting drug use (within the last 6 months) or receiving opioid substitution therapy (OST).

In addition to the above interventions, participants will complete a survey. They will also be invited to provide consent to link data with routinely collected data from a range of population databases and registers.

Participant recruitment will take place in public and private drug treatment clinics, high case-load GPs, and NSP programmes.

A sub study will be included in ETHOS ENGAGE. As part of this sub-study, 550 participants will be invited to provide a sample of blood collected via venepuncture, which will be used to evaluate simplified HCV diagnostic assays on finger-stick and DBS samples to diagnose chronic HCV infection.

Part II: Qualitative Interviews Policy makers, clinicians and patients from selected clinics will be interviewed to examine barriers and facilitators to HCV care.

Part III: HCV toolkit, education and training A HCV education and training program (including HCV tool-kit) will be developed in collaboration with ASHM, based on learnings generated through ETHOS ENGAGE and the qualitative interviews, to enhance workforce development and improve HCV care in drug treatment clinics and needles and syringe programmes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has voluntarily signed the informed consent form;
* 18 years of age or older;
* History of injecting drug use*;
* Recent injecting drug use (previous six months) or currently receiving OST*.

  * These criteria will not apply for recruitment from residential rehabilitation centres

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants commencing anti-HCV treatment | Every year post enrolment for up to 3 years
  Evaluation of number of participants commencing anti-HCV treatment

CONTACTS AND LOCATIONS:
Locations (29):
- Australia (29):
  - NSLHD Brookvale Community Health Centre, Brookvale, New South Wales
  - Coopers Cottage, Campbelltown Drug Health Services, Campbelltown, New South Wales
  - HNELHD Drug and Alcohol Clinical Services Cessnock, Cessnock, New South Wales
  - MNCLHD Coffs Harbour Alcohol and Other Drug Services, Coffs Harbour, New South Wales
  - Rankin Court Treatment Centre, Darlinghurst, New South Wales
  - NNSWLHD Grafton Alcohol and Other Drug Services, Grafton, New South Wales
  - NBMLHD Drug & Alcohol Services Katoomba, Katoomba, New South Wales
  - MNCLHD Kempsey Alcohol and Other Drug Services, Kempsey, New South Wales
  - NBMLHD Drug & Alcohol Services Nepean, Kingswood, New South Wales
  - NNSWLHD Lismore (Riverlands) Alcohol and Other Drug Services, Lismore, New South Wales
  - NBMLHD Drug & Alcohol Services Lithgow, Lithgow, New South Wales
  - Liverpool Opioid Treatment Program, Liverpool, New South Wales
  - WSLHD Mount Druitt Drug Health OST Clinic, Mount Druitt, New South Wales
  - HNELHD Drug and Alcohol Clinical Services Newcastle, Newcastle, New South Wales
  - Lawrence Avenue Methadone Program (LAMP), Nowra, New South Wales
  - WSLHD Fleet Street Drug Health OST Clinic, Parramatta, New South Wales
  - MNCLHD Port Macquarie Alcohol and Other Drug Services, Port Macquarie, New South Wales
  - NSLHD Herbert Street Clinic, Saint Leonards, New South Wales
  - HNELHD Drug and Alcohol Clinical Services Tamworth, Tamworth, New South Wales
  - HNELHD Drug and Alcohol Clinical Services Taree, Taree, New South Wales
  - NNSWLHD Tweed Heads Alcohol and Other Drug Services, Tweed Heads, New South Wales
  - The Orana Centre, Wollongong, New South Wales
  - Roma Street Clinic, Brisbane, Queensland
  - Youthlink, Cairns, Queensland
  - Northern Drug and Alcohol Services South Australia (DASSA), Elizabeth, South Australia
  - Central Drug and Alcohol Services South Australia (DASSA), Stepney, South Australia
  - Next Step Fremantle, Fremantle, Western Australia
  - Next Step Joondalup, Joondalup, Western Australia
  - Next Step East Perth, Perth, Western Australia